CLINICAL TRIAL: NCT04581707
Title: Evaluation of Surgical Therapy of Vertebral Compression Fractures With the Kyphoplasty Single Balloon Catheter Allevo (Joline®) and the Quattroplasty Double Balloon Catheter Stop'n GO (Joline®) With BonOs® Inject Bone Cement
Brief Title: Performance and Safety of Joline® Kyphoplasty Single Balloon Catheter Allevo vs. Quattroplasty Double-Balloon Catheter Stop'n GO With BonOs® Inject Bone Cement
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital Tuebingen (Other)
Responsible Party: Principal Investigator, Lisanne Exner, Medical assistant, University Hospital Tuebingen
Other Study IDs: JO-2020Kypho
Record Dates: First submitted 2020-09-18; First posted 2020-10-09 (Actual); Last update posted 2021-01-19 (Actual); Status verified 2021-01

CONDITIONS: Vertebral Compression Fracture
Keywords: Vertebral augmentation; Balloon kyphoplasty systems; Bone cement

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Kyphoplasty Single Balloon Catheter Allevo
  Interventions: Device: Kyphoplasty Single Balloon Catheter Allevo
- Quattroplasty Double Balloon Catheter Stop'n GO
  Interventions: Device: Quattroplasty Double Balloon Catheter Stop'n GO

INTERVENTIONS:
Device: Kyphoplasty Single Balloon Catheter Allevo — Vertebral compression fractures treated with Kyphoplasty Single Balloon Catheter Allevo (Joline®) and BonOs® Inject bone cement
  Groups: Kyphoplasty Single Balloon Catheter Allevo
Device: Quattroplasty Double Balloon Catheter Stop'n GO — Vertebral compression fractures treated with Stop'n GO double balloon kyphoplasty system (Joline®) and BonOs® Inject bone cement
  Groups: Quattroplasty Double Balloon Catheter Stop'n GO

SUMMARY:
The purpose of this study is to assess the performance and safety of two balloon kyphoplasty systems (Joline®), the single balloon catheter Allevo and Quattroplasty double balloon catheter Stop'n Go, using BonOs® Inject bone cement for treatment of Vertebral Compression Fractures.

DETAILED DESCRIPTION:
Vertebral compression fracture (VCF) is a very common medical problem and describes the collapse of a vertebral body (VB) in the spine. VCF can lead to severe pain, decreased physical function, spinal deformity and in rare cases thoracic or abdominal wall deformities, that can impair pulmonary and gastrointestinal function. A VCF can occur in patients with healthy spines upon severe trauma, in patients suffering from osteoporosis or in patients with metastatic tumors.

Currently available therapy for VCF includes medical management, surgical treatments and vertebral augmentation (VA). Medical management consists of bed rest followed by early mobilization and analgesic medications. Surgical options include spinal stabilization with rods and screws. VA procedures attempt to stabilize the spine and reduce vertical compression by adding material to the spine.

Kyphoplasty is a commonly performed VA procedure. In kyphoplasty, a surgical instrument is used to reduce the collapsed VB towards its original shape. Reduction of the fractured VB is thought to be beneficial since (1) it may reduce anterior directed compressive forces resulting from kyphosis of the spine due to the fracture, and (2) it may reduce some physiologic abnormalities due to kyphosis, such as restrictive lung disease or abdominal compression. After fracture reduction, bone cement is placed in the VB to stabilize the reduction. Fracture reduction follows the orthopedic general principles of fracture repair: reduction and stabilization.

Primary objective of this observational study is to compare the effectiveness of the Quattroplasty double balloon catheter Stop'n GO (Joline®) with the Kyphoplasty single balloon catheter Allevo (Joline®) combined with BonOs® Inject bone cement for use in VCF reduction, to confirm the performance of those two devices and to investigate potential major adverse events associated with the use of the device in patients treated in a controlled setting when used according to the IFU. Secondary objective is to compare the safety of the Quattroplasty double balloon catheter Stop'n GO (Joline®) with the Kyphoplasty single balloon catheter Allevo (Joline®) combined with BonOs® Inject bone cement.

ELIGIBILITY:
Inclusion Criteria:

* patients aged ≥18 years
* 1-3 painful VCF(s), of which at least 1 meets the following criteria:

  * VCF between T7 and L5
  * Fracture age <3 months
  * VCF shows hyperintense signal on STIR or T2 sequence MRI.
* Investigator estimates that target VB(s) is/ are suitable for Quattroplasty double balloon catheter or Kyphoplasty single balloon catheter (e.g. appropriate pedicle diameter, no cortical bone protruding into the spinal canal).
* Patient has an ODI score of 30% or more.
* Patient is willing and able to comply with study requirements.
* Patient signs informed consent form.
* Women who are post-menopausal, surgically sterile or on contraceptives and agree to remain on contraceptives for the duration of their study participation and agree not to become pregnant during the study.

Exclusion Criteria:

* Segmental kyphosis of target VB of >30°
* Pre-existing or clinically unstable neurologic deficit
* Any physical exam evidence of myelopathy or radiculopathy
* Not able to walk without assistance prior to fractures
* Any radiographic evidence of pedicle fracture or interspinous-process widening
* Spondylolisthesis >grade 1 at target VB(s)
* History of spine surgery, including prior vertebral augmentation, during the last year
* Any underlying systemic bone disease other than osteoporosis (e.g. osteomalacia, osteogenesis imperfect, etc.)
* Irreversible coagulopathy and/or taking peri-operatively warfarin (Coumadin) or other anticoagulant
* Pregnancy and nursing
* Pain due to any other condition that requires daily narcotic medication
* Disabling back pain due to causes other than acute fracture
* History of intolerance, or allergic reaction to titanium or acrylic compounds
* Active systemic or local infection at baseline
* Severe cardiopulmonary disease (e.g. stage IV heart failure, severe chronic obstructive pulmonary disease)
* Any other medical illness or condition that, in the investigator's opinion, is likely to impair long-term follow-up (e.g. cancer) or greatly increase the risk of surgery
* Any evidence of substance abuse
* The patient is on long-term steroid therapy (steroid dose 30 mg/day for >3 months)
* The patient is known to be involved in medical litigation including Workmen's compensation.
* Patient with contraindication for MRI including but not limited to patients with contraindications for general anesthesia (surgeon expertise)
* Patient who is contraindicated for the use of PMMA cement
* Patients who belong to a vulnerable population or that are not able to sign the informed consent form.
* Patients where the VCF was treated in combination with fusion.
* Patients with any contraindication according to the IFU

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing or patients who have already undergone percutaneous balloon kyphoplasty for treatment of Vertebral Compression Fractures as indicated in the Instructions for use of the investigational devices.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2020-03-01 (Actual); Primary Completion 2021-06 (Estimated); Study Completion 2021-10 (Estimated)

PRIMARY OUTCOMES:
Change in vertebral body height | pre-operative, 5 days and 3 months post-operatively
  Change in vertebral body height
Change in Visual Analog Scale (VAS) of subjective pain | pre-operation, 5 days and 3 months post-operation
  The Visual Analog Scale (VAS) is a measure for pain intensity. The score of the sclae ranges from 0 for "no pain" to 10 for "worst imaginable pain". Patients will report their pain at baseline and at 2 dedicated periods to assess change in pain intensity.
Change in functional disability | pre-operation, 5 days and 3 months post-operation
  The Oswestry Disability Index (ODI) is used to assess functional disability. The questionnaire consists of 10 items with each item having 6 statements. All scores are summed, then multiplied by two to obtain the index (range from 0 to 100) with higher score indicating greater disability.

SECONDARY OUTCOMES:
Safety Outcomes: Occurence of adverse events and complications | during procedure, 5 days and 3 months post-operation
  Occurence of adverse events and complications

CONTACTS AND LOCATIONS:
Overall Officials: Lisanne Exner, Principal Investigator — University Hopsital for Orthopedics Tuebingen
Locations (1):
- University Hospital for Orthopedics Tuebingen, Tübingen, Germany

IPD SHARING:
Plan to Share IPD: No